CLINICAL TRIAL: NCT01293422
Title: PXR-aktivaation Vaikutukset Sokeri-, Kolesteroli- ja Hormonitasapainoon
Brief Title: Effects of Pregnane X Receptor (PXR) Activation on Human Glucose, Lipid and Hormone Homeostasis
Acronym: Rifa-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Rifa-2; 2010-023662-47 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Glucose Metabolism
Keywords: PXR, glucose, cholesterol
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifampicin (Experimental)
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — Rifampicin 600 mg daily for a week
  Other Names: Rimapen, ATC J04AB02

SUMMARY:
This clinical trial is designed to study the effects of pregnane X receptor activator rifampicin on the glucose, lipid and hormone homeostasis in healthy volunteers. The main hypothesis is that rifampicin raises postprandial glucose studied with oral glucose tolerance test. The study is a non-randomized, one-phase, open-label trial. Twelve subjects will be given 600 mg of rifampicin a day for a week. The main outcome measures are the changes in the glucose and insulin levels during oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age 18-45 years
* Body mass index 19-28

Exclusion Criteria:

* Any continuous medication
* Any significant disease
* Allergy to rifampicin
* Pregnancy and breast feeding
* Fear of needles and previous difficult blood samplings
* Substance abuse
* Participation in another clinical drug trial within 1 month of enrollment
* Use of soft contact lenses

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Glucose levels during oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Rahunen R, Kummu O, Koivukangas V, Hautajarvi H, Hakkola J, Rysa J, Hukkanen J. Pregnane X Receptor-4beta-Hydroxycholesterol Axis in the Regulation of Overweight- and Obesity-Induced Hypertension. J Am Heart Assoc. 2022 Mar 15;11(6):e023492. doi: 10.1161/JAHA.121.023492. Epub 2022 Mar 1. PMID 35229613